CLINICAL TRIAL: NCT05406687
Title: Cancer Prevention and Early Detection Among the Homeless Population in Europe: Co-adapting and Implementing the Health Navigator Model
Brief Title: Cancer Prevention and Early Detection Among the Homeless Population: The Health Navigator Model
Acronym: CANCERLESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Valencia (Other); Senior Europa Sociedad Limitada (Unknown); Ministry of Social Policies and Family, Spain (Unknown); Servicio Madrileño de Salud, Madrid, Spain (Other); International Foundation for Integrated Care (Unknown); Programs of Development, Social Support and Medical Cooperation Association (Unknown); European Federation of National Organisations working with the Homeless (Unknown); Prolepsis Institute for Preventive, Environmental and Occupational Medicine (Other); Anglia Ruskin University (Other); Universitat Politècnica de València (Other)
Responsible Party: Principal Investigator, Igor Grabovac, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 965351
Record Dates: First submitted 2022-05-19; First posted 2022-06-06 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: Europe; Cancer; Cancer prevention; Primary care; Co-designed intervention; Implementation science; Homelessness; Homeless population; Longitudinal; Person-centered
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People experiencing homelessness (Other): All homeless adults, aged 18 years and over, who visit the CANCERLESS pilot sites will be asked to participate (convenience sampling). We define individuals as being homeless if they fall under one of the categories listed in the European typology of homelessness and housing exclusion.
  Interventions: Other: Health Navigator Model

INTERVENTIONS:
Other: Health Navigator Model — The Health Navigator Model will be a longitudinal, person-centered and community-based intervention focused on addressing both primary and secondary cancer prevention, as well as reducing wider barriers to healthcare. Health Navigators (HNs) will be professionals who have a background in social care and an understanding of the local user population, and will be embedded in settings familiar and accessible to people experiencing homelessness. The primary aspects of the HN role will be to identify the health needs and barriers of users, promote cancer awareness and education, facilitate timely access to healthcare services and cancer screening, provide practical assistance, delivered through regular in-person meetings, and utilize wider stakeholders, including healthcare professionals, to deliver the intervention. A comprehensive training package will be delivered to the HNs, covering population specific knowledge, interpersonal skills, cancer education and local resources.

SUMMARY:
Prevention and early detection are key for the decrease of cancer-related mortality. However, socially deprived population groups don't have the privilege of unburdened access to the healthcare system. The EU-funded CANCERLESS project aims to develop an evidence-based, patient-centred innovation that reinforces patients through health education and social support and fosters timely access to primary and secondary prevention services. Based on the combination of the tested Patient Navigator Model and the Patient Empowerment Model, CANCERLESS will develop the Health Navigator Model for Europe, addressed to the underserved population.

DETAILED DESCRIPTION:
Homeless individuals have higher prevalence of adverse health outcomes (infectious diseases, substance-related disorders, etc.) and premature mortality compared to the general population, with cancer being the second most common cause of death. In most cases, people experiencing homelessness experience significant barriers or do not have access to community health services, including access to primary and secondary prevention services and programs. Cancer prevention and early detection among the homeless population in Europe: Co-adapting and implementing the Health Navigator Model - The CANCERLESS project is a Horizon 2020 financed project aiming to adapt a novel, evidence based and person-centered model to address this underserved population and eliminate barriers to access primary and secondary preventive services.

The Health Navigator Model (HNM), a person-centered intervention co-designed during the first part of the project, will address the growing health and social disparities in the homeless population and promote timely access to cancer prevention and screening services. Therefore, the aim of this longitudinal, person-centered, and community-based intervention study is to pilot test the HNM by investigating a cohort of individuals experiencing homelessness in pilot-sites in Austria, Greece, Spain and the United Kingdom. Our study will assess whether the HNM intervention can improve the delivery of evidence of community-based primary and secondary cancer preventive care for the homeless population. The HNM will be conducted over a set time frame, with active participation being individually tailored to the needs of participants, within an overall period of 18 months. Evaluation will be performed at baseline and at three further evaluation points to assess the outcomes of the intervention. Adult individuals experiencing homelessness (as defined by the European Topology of Homelessness and Housing Exclusion) will be asked to participate during their visits to the pilot sites of cooperating facilities (non-governmental organizations offering free medical care, or social service institutions) after assessing eligibility criteria.

The study utilizes both a qualitative and quantitative methodology which will allow us to conduct both exploratory and confirmatory research and thus, gain a deeper comprehension of the impact of the HNM intervention on overall participation of homeless individuals in primary and secondary cancer preventive programs.

The project has been funded by the HORIZON 2020 program of the European Commission under the topic: "H2020-SC1-2020-Single-Stage-RTD - Call for proposals on the prevention and/or early diagnosis of cancer" and is coordinated by the Medical University of Vienna.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* No diagnosed cancer
* Any category of the European Typology of Homelessness and housing exclusion applies
* Sufficient knowledge of language

Exclusion Criteria:

* Persons who cannot give consent due to diminished capacity
* Persons who do not provide informed consent
* Known cancer diagnosis
* Cancer survivorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Clinical utility/effectiveness | 18 months
  The first objective of the CANCERLESS evaluation is to determine the clinical utility/effectiveness of the Health Navigator Model intervention on the health promotion and cancer primary and secondary prevention among people experiencing homelessness. Effectiveness refers to the likelihood that a certain protocol (in this case the Health Navigator Model) will benefit users in a certain population (in this case people experiencing homelessness) by resulting in an improved health outcome. Therefore, the clinical utility/effectiveness evaluation will include the assessment of the differences between baseline and follow-up measurements, especially on health outcomes among those people experiencing homelessness that participate in the project.
Cost-effectiveness and cost-utility | 18 months
  In addition to the effectiveness evaluation, CANCERLESS aims to determine the cost-effectiveness and cost-utility of the Health Navigator Model implementation. In regard to the cost-effectiveness and cost-utility analyses, these refer to the degree to which the application of the Health Navigator Model for prevention of cancer among the homeless population is effective or productive in relation to its cost. To conduct this economic evaluation, health outcomes, such as quality of life, and the cost required to achieve the expected health and well-being results providing the Health Navigator Model will be analyzed. This analysis will be based on the data collected on health outcomes and costs (healthcare costs and cancer costs and burden) within the project.
Facilitators and barriers for the Health Navigator Model implementation | 18 months
  Finally, the third objective is aimed at identifying factors acting as facilitators and barriers for an effective and successful implementation of the Health Navigator Model under the CANCERLESS project. To this aim, not only patients or users' experiences will be taken into account, but also the feedback from navigators and multidisciplinary teams participating in CANCERLESS project. Also, analyses of the differences between baseline and follow-up measurements will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Grabovac, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (18):
- AmberMed, Vienna, Austria
- Greece (3):
  - PRAKSIS Open Day Center for Homeless Athens, Athens, Attica
  - PRAKSIS Open Day Center for Homeless Piraeus, Piraeus, Attica
  - PRAKSIS Community Center, Sepolia, Attica
- Spain (12):
  - Centro de Salud Segre, Madrid
  - Centro de Salud Segovia, Madrid
  - Samur Social, Madrid
  - Centro de Salud Casa de Campo, Madrid
  - Centro de Salud Cortes, Madrid
  - Centro de Salud Justicia, Madrid
  - Centro de Salud Benita de Ávila, Madrid
  - Centro de Salud Las Águilas, Madrid
  - Shelter el Pinar, Madrid
  - Shelter San Isidro, Madrid
  - Shelter San Juan de Dios, Madrid
  - Women's centre Beatriz Galindo, Madrid
- United Kingdom (2):
  - The Purfleet Trust - Pathway House, Kings Lynn, Norfolk
  - Dibden Road Hostel (Part of St Martins Housing Trust), Norwich, Norfolk

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised and limited data set may be given to other researchers upon request from the principal investigator, following compliance of the Data Security Department of the Medical University of Vienna.

REFERENCES:
- [Derived] Carmichael C, Schiffler T, Smith L, Moudatsou M, Tabaki I, Donate-Martinez A, Alhambra-Borras T, Kouvari M, Karnaki P, Gil-Salmeron A, Grabovac I. Barriers and facilitators to health care access for people experiencing homelessness in four European countries: an exploratory qualitative study. Int J Equity Health. 2023 Oct 6;22(1):206. doi: 10.1186/s12939-023-02011-4. PMID 37803317
- See also: Related Info — https://cordis.europa.eu/project/id/965351